CLINICAL TRIAL: NCT03085108
Title: Validation and Mapping of the Suicide Ideation and Behavior Assessment Tool in Subjects at Various Levels of Risk for Suicide
Brief Title: A Study to Assess the Validation and Mapping of the Suicide Ideation and Behavior Assessment
Status: Completed | Type: Observational
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108248; 54135419SUI0001 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2017-03-14; First posted 2017-03-21 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Suicidality
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SIBAT, the S-STS CMCM, and the C-SSRS + CGI-SS-R: Participants randomized to Cohort A will be consented for video-recorded interviews on 3 distinct suicide assessment instruments (the Suicide Ideation and Behavior Assessment Tool [SIBAT], the Sheehan-Suicidality Tracking Scale Clinically Meaningful Change Measure [S-STS CMCM] and the Columbia-Suicide Severity Rating Scale [C-SSRS] + Clinical Global Impression of Severity of Suicidality (Revised) [CGI SS-R]). These participants will be interviewed 3 times within the single study visit by 3 different trained clinical raters, using semi-structured interviews that have been developed for each of the 3 suicide assessment instruments.
  Interventions: Other: No Intervention
- SIBAT: Participants who are not videotaped for the 3 interviews will only be assessed by SIBAT.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The main purpose of this cross-sectional study is to generate data to support the psychometric properties of the Suicide Ideation and Behavior Assessment Tool (SIBAT) and validate its use in participants at imminent risk of suicide.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be able to speak, read, and write English sufficiently well to complete consent process and self-administer study questionnaires
* Each participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of the interviews and, when applicable, the videotaping required for the study and are willing to participate in the study. Adolescents (minors) who in the judgment of the investigator are capable of understanding the nature of the study can be enrolled only after obtaining consent of a legally acceptable representative. Assent must be obtained from any participating adolescents (minors)
* Each participant or legally acceptable representative must check a separate box on the consent form if he or she agrees to have interviews video-recorded. Participants who do not consent to video recording will only be administered the SIBAT

Exclusion Criteria:

- Participant has any clinically relevant physical or mental conditions including, but not limited to vision problems, physical disability, severe mental illness, or cognitive impairment (such as from acute intoxication or dementia) which, in the opinion of the investigator, would interfere with ability to complete the study interviews

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants in this study will be selected from emergency room, acute inpatient psychiatric hospital unit, or psychiatry clinical research office settings. Participants who agree to be interviewed regarding their symptoms of suicidality will be screened and selected if they meet selection criteria for this study. Participants with various levels of suicidality will be included based on the severity of their suicidality assessed globally (without extensive interview).
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression of Severity of Suicidality (Revised) (CGI-SS-R) | Day 1
  The Clinical Global Impression - Severity of Suicidality - Revised (CGI-SS-R) was derived from the Clinical Global Impression Severity Scale (CGI-S), a global rating scale that gives an overall measure of the severity of a participants illness. The CGI-SS-R rating is scored on a 7-point scale from 0 (normal, not at all suicidal) to 6 (among the most extremely suicidal participants).
Clinical Global Impression of Imminent Suicide Risk (CGI-SR-I) | Day 1
  CGI-SR-I describes aspects of participant's suicidal thinking, behavior and related contributory/protective factors, what is best clinical judgment of participant's imminent risk for suicide within the next 7 days. Scale indicates: 0 (No imminent suicide risk), 1 (Minimal imminent), 2 (Mild imminent), 3 (Moderate imminent), 4 (Marked imminent), 5 (Severely imminent), 6 (Extreme imminent).
Clinical Global Impression of Long Term Suicide Risk (CGI-SR-LT) | Day 1
  CGI-SR-I describes aspects of participant's suicidal thinking, behavior and related contributory/protective factors, what is best clinical judgment of participant's imminent risk for suicide (that is, they will likely end their life by suicide sometime in the future). Scale indicates : 0 (No suicide risk in the long term), 1 (Minimal suicide risk), 2 (Mild suicide risk), 3 (Moderate suicide risk), 4 (Marked suicide risk), 5 (Serious suicide risk), 6 (Extreme risk).
Frequency of Suicidal Thinking (FoST) | Day 1
  Frequency of Suicidal Thinking describes the clinician determined estimate of the frequency of the participant's suicidal thinking (The FoST rating is scored on a 6-point Likert scale : 0 (Never), 1 (Rarely), 2 (Sometimes), 3 (Often), 4 (Most of the time), 5 (All of the time).
Columbia-Suicide Severity Rating Scale [C-SSRS]) | Day 1
  C-SSRS is a clinician rated assessment of suicidal behavior and / or intent. Scale consists of 28 items in 4 sections: suicide behavior, actual attempts, suicidal ideation, and intensity of ideation. Suicidal ideation consists of 5 'yes/no' items: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intention to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent. Only items with yes responses are listed. Worsening of suicidal ideation was an increase in severity of suicidal ideation from baseline.
Sheehan-Suicidality Tracking Scale Clinically Meaningful Change Measure [S-STS CMCM] | Day 1
  The S-STS CMCM is a multi-item scale that can be administered either by a clinician or patient through self-report. Each item in the S-STS CMCM patient self-report suicide phenomena section (14 items) is scored on a 5-point Likert scale : 0 (not at all), 1 (a little), 2 (moderately), 3 (very), and 4 (extremely).

SECONDARY OUTCOMES:
Suicide Ideation and Behavior Assessment-My Risk/Protective Factors | Day 1
  Patient-reported dynamic suicide risk and protective characteristics (My Risk/Protective Factors) will be assessed based on Suicide Ideation and Behavior Assessment Tool (SIBAT) with up to 31 items that best describes how participant have acted or felt in the past 7 days in terms of responses (Never, Rarely, Sometimes, Often, Most of the time, All the time). This best describes how participants are thinking or feeling right now in terms of Strongly Disagree, Disagree, Slightly Disagree, Slightly agree, Agree, Strongly Agree.
Suicide Ideation and Behavior Assessment: My Current Thinking | Day 1
  Patient-reported current suicide ideation (My current thinking) will be assessed based on SIBAT with 48 items. The best describes how participants are thinking or feeling right now in terms of Strongly Disagree, Disagree, Slightly Disagree, Slightly agree, Agree, Strongly Agree.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - CNS Network, Garden Grove, California
  - Rutgers University, Piscataway, New Jersey
  - University of Cincinnati, Cincinnati, Ohio